CLINICAL TRIAL: NCT06941987
Title: Evaluate the Clinical Feasibility of a Novel Neoantigen-Reactive CD8+ T Cell (NART) Detection Technology for Postoperative MRD Surveillance of Pancreatic Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZSPAC-11
Record Dates: First submitted 2025-04-12; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-03

CONDITIONS: Minimal Residual Disease; Pancreatic Cancer Resectable
MeSH Terms: conditions — Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the diagnostic performance of a novel Neoantigen-Reactive CD8+ T cell (NART) technology detecting minimal residual disease (MRD) in postoperative surveillance of pancreatic cancer. The main question it aims to answer is: Is NART a sensitive and accurate detection for MRD? Participants are required to undergo periodic blood sampling and imaging examinations as the protocol specifies.

ELIGIBILITY:
Inclusion Criteria:

* age >18
* Assessd as resectable PDAC before surgical procedure
* Voluntary to donate tumor samples resected in curative surgery for PDAC
* Voluntary to participate in the radiological evaluation, tests of serum tumor markers, and the collection of MRD samples according to the study protocol
* ECOG state (PS) grades ≤ 2
* Voluntary to sign informed consent and adhering to the requirements and limitations outlined by lCD and this protocol
* Confimed as pancreatic ductal adenocarcinoma by pathology
* RO or R1 resection
* Clinically evalutated eligible for adjuvant therapy
* Tumor tissue samples meet the requirements of whole exome sequencing (WES)

Exclusion Criteria:

* Preoperative imaging examinations show distant metastasis
* Have received neoadjuvant therapy
* Have any other active malignancy within 5 years before enrollment, or have any other indolent cancers that did not interfere with the primary cancer assessment in the study without prior approval from the research committee
* With other physical or mental conditions that may increase the risk of study participation or (in the investigator's judgment) may make the subject ineligible for study participation, including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormalities
* Have participated in other interventional or observational clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receive radical resection without naoadjuvant therapy and diganosed pancreatic ductal adenocarcinoma pathologically are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2025-10-20 (Estimated); Study Completion 2027-10-20 (Estimated)

PRIMARY OUTCOMES:
The correlation between NART detection and recurrence-free survival | From date of surgery until the date of diagnosis of local or metastatic recurrence, assessed 3 months thereafter up to 60 months

SECONDARY OUTCOMES:
The correlation between conventional ct-DNA test and RFS | From date of surgery until the date of diagnosis of local or metastatic recurrence, assessed 3 months thereafter up to 60 months
The correlation between serum markers and RFS | From date of surgery until the date of diagnosis of local or metastatic recurrence, assessed 3 months thereafter up to 60 months
The correlation between NART detection and overall survival (OS) | From date of surgery until the date of death, assessed 3 months thereafter up to 60 months
The correlation between conventional ct-DNA test and OS | From date of surgery until the date of death, assessed 3 months thereafter up to 60 months
The correlation between serum markers and OS | From date of surgery until the date of death, assessed 3 months thereafter up to 60 months
The diagnostic performance of NART detection | From the date of first enrollment until the study completion, an average of 30 months.
  Evaluation index of diagnostic performance include: sensitivity, specificity, positive predictive value, negative predictive value and lead time advantages over radiological recurrence manifestations. Sensitivity is defined as the proportion of subjects who tested positive for MRD/elevated serum tumor markers at or before recurrence confirmed by clinical imaging. Specificity was defined as the proportion of subjects who tested negative for MRD/normal serum tumor markers at or before clinical imaging confirmation of relapse. Positive Predictive Value (PPV) and Negative Predictive Value (NPV) are defined as the proportion of subjects testing MRD-positive/negative who are clinically confirmed to relapse/remain relapse-free, respectively. Lead time is defined as the time interval from MRD positivity or serum tumor marker elevation to imaging-confirmed clinical relapse.
The diagnostic performance of conventional ct-DNA test. | From the date of first enrollment until the study completion, an average of 30 months.
  Evaluation index of diagnostic performance include: sensitivity, specificity, positive predictive value, negative predictive value and lead time advantages over radiological recurrence manifestations. Sensitivity is defined as the proportion of subjects who tested positive for MRD/elevated serum tumor markers at or before recurrence confirmed by clinical imaging. Specificity was defined as the proportion of subjects who tested negative for MRD/normal serum tumor markers at or before clinical imaging confirmation of relapse. Positive Predictive Value (PPV) and Negative Predictive Value (NPV) are defined as the proportion of subjects testing MRD-positive/negative who are clinically confirmed to relapse/remain relapse-free, respectively. Lead time is defined as the time interval from MRD positivity or serum tumor marker elevation to imaging-confirmed clinical relapse.
The diagnostic performance of serum markers. | From the date of first enrollment until the study completion, an average of 30 months.
  Evaluation index of diagnostic performance include: sensitivity, specificity, positive predictive value, negative predictive value and lead time advantages over radiological recurrence manifestations. Sensitivity is defined as the proportion of subjects who tested positive for MRD/elevated serum tumor markers at or before recurrence confirmed by clinical imaging. Specificity was defined as the proportion of subjects who tested negative for MRD/normal serum tumor markers at or before clinical imaging confirmation of relapse. Positive Predictive Value (PPV) and Negative Predictive Value (NPV) are defined as the proportion of subjects testing MRD-positive/negative who are clinically confirmed to relapse/remain relapse-free, respectively. Lead time is defined as the time interval from MRD positivity or serum tumor marker elevation to imaging-confirmed clinical relapse.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai, China

IPD SHARING:
Plan to Share IPD: No